CLINICAL TRIAL: NCT06162260
Title: Analyse Des Facteurs de Risque Pour la réintégration Non planifiée Post-opératoire de Patients transplantés du Foie Chez l'Enfant
Brief Title: Unplanned ICU Readmission for Pediatric Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: gaoleiqing
Record Dates: First submitted 2023-12-01; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Liver Transplantation
Keywords: readdmission;ICU;transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observation group: (1) Liver transplantation was performed between January 1, 2019 and December 31, 2019; (2) Age < 18 years; (3) The patient was admitted to ICU for the first time due to postoperative monitoring after liver transplantation; (4) Survival on first transfer from ICU.
  Interventions: Procedure: ICU readmission
- matched group: (1) Liver transplantation was performed between January 1, 2019 and December 31, 2019; (2) Age < 18 years; (3) The patient was admitted to ICU for the first time due to postoperative monitoring after liver transplantation; (4) survive the first transfer from ICU; (5) No ICU re-entry occurred in the same hospitalization period after liver transplantation.

INTERVENTIONS:
Procedure: ICU readmission — Children who underwent liver transplantation at Renji Hospital, Shanghai Jiao Tong University School of Medicine from January 1, 2018 to December 31, 2021 and were transferred out of ICU for the first time during the same hospitalization cycle.
  Groups: observation group

SUMMARY:
To explore the risk factors of unplanned return to Intensive Care Unit (ICU) in pediatric liver transplant recipients, and to provide data support for the transfer of pediatric liver transplant recipients from ICU after surgery, so as to avoid unplanned ICU return and reduce the mortality of patients during hospitalization.

DETAILED DESCRIPTION:
In recent years, with the progress of medical level, pediatric liver transplantation has been used in a variety of pediatric end-stage liver diseases, such as intrahepatic cholestasis, metabolic diseases, acute liver failure, liver tumors and other diseases. It is the only effective way to treat pediatric end-stage liver diseases. The maturity of surgical techniques and the application of immunosuppressants have greatly improved the overall survival rate of children after liver transplantation. In some developed countries, the 1-year and 5-year survival rates of children after liver transplantation can reach more than 80%. Pediatric liver transplantation is difficult, and the postoperative condition is complicated and changes rapidly, which requires Intensive Care Unit (ICU) for intensive monitoring. However, unplanned reentry to the ICU occurs in some pediatric liver transplant recipients who have been transferred out of the ICU and need to be transferred again because of a change in their condition. Unplanned ICU return leads to increased mortality, longer hospital stay, and higher hospital costs. For example, Rosenberg et al. [5] reported that the comprehensive ICU re-entry rate was 4-14% (average 7%), the average length of stay was more than twice that of non-re-entrants, and the mortality rate was 2-10 times that of non-re-entrants. Kramer et al. [8] analyzed 229375 patients in 97 intensive care units from 2001 to 2009, and the re-entry rate was 6.1%. The average length of stay of the re-entry patients was 2.5 times higher than that of the non-re-entry patients, and the mortality rate was 4 times higher than that of the non-re-entry patients. Therefore, unplanned ICU re-entry is a rare but serious event, which has important clinical significance for the study of unplanned ICU re-entry.

There are significant differences in ICU re-entry rates among liver transplant recipients in different studies. Young Gon Son et al. reported that 5.8% (68 patients /1181 patients) of the enrolled patients underwent ICU re-entry after liver transplantation. A case-control study at a Canadian medical center showed that 14% of 369 patients who received liver transplants at the center between 2005 and 2012 had ICU re-entry; They had a longer first hospital stay (P<0.001) and a lower cumulative survival rate of 1 month to 2 years (P<0.001). The study by Mark et al. showed that ICU re-entry occurred in 34% of 167 liver transplant recipients. Several studies of risk factors for ICU return after liver transplantation have also shown mixed results. For example, Levy et al. showed that older age and more intraoperative blood transfusion in liver transplant recipients were positively associated with ICU return. Filipe et al. showed that more than 20 breaths per minute at ICU discharge after liver transplantation was an independent risk factor for ICU return during the same hospitalization. At present, studies on ICU re-entry rate and risk factors after liver transplantation mostly focus on adult liver transplant recipients. There are no reports on risk factors for ICU return after liver transplantation in children. Some reports of PICU's return were found. For example, Angela S statistically analyzed 117,923 children admitted to 73 PICUs from 2005 to 2008. The ICU re-entry rate was 3.7%, of which 38%(1.4%) occurred early (ICU re-entry within 48 hours). Patient characteristics strongly associated with an increased risk of early readmission included age < 6 months, acute respiratory and renal disease, and underlying chronic conditions such as liver disease, bone marrow transplantation, and airway stenosis. Afrothite Kotsakis's study showed that younger age, lower body weight, longer first ICU stay, and non-target time transfer (06:00-11:59) were among the factors affecting children's ICU return. Can these conditions and risk factors for PICU re-entry and ICU re-entry in adult liver transplant recipients be applied to analyze ICU re-entry in pediatric liver transplant recipients? We don't know. Because there is a significant physiological difference between adults and children, liver transplantation is difficult to apply PICU reentry cause analysis due to the difficulty of operation and the uniqueness of immunosuppressive therapy. In other words, risk factors for postoperative ICU return in pediatric liver transplant recipients may differ from those in adult liver transplant recipients and other children. Therefore, a separate analysis of risk factors for unplanned ICU return after liver transplantation in children is necessary.

ELIGIBILITY:
Inclusion Criteria:

* (1) Liver transplantation was performed from January, 2018 to December, 31, 2021.21;
* (2) Age < 18 years;
* (3) The patient was admitted to ICU for the first time due to postoperative monitoring after liver transplantation;
* (4) Survival on first transfer from ICU.

Exclusion Criteria:

* (1) Death during ICU stay after liver transplantation;
* (2) non-first-time recipients of liver transplantation;
* (3) Patients with complex conditions who were transferred to ICU for life support (such as mechanical ventilation, CRRT, etc.) before operation;
* (4) Patients admitted to ICU by appointment for surgical reasons.
* (5) Patients forcibly transferred from ICU.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who underwent liver transplantation at Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine from Jan 1, 2018 to Dec 31, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 1575 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-29 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Unplanned return to the ICU | 01/01/2018-31/12/2021
  ICU re-entry occurred within the same hospital cycle after the first ICU transfer after liver transplantation

IPD SHARING:
Plan to Share IPD: Undecided